CLINICAL TRIAL: NCT01873274
Title: Comparative Study of Three Delivery Systems of Menaquinone-7
Brief Title: Comparative Study Menaquinone-7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-3-009
Record Dates: First submitted 2013-05-30; First posted 2013-06-10 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- basic yogurt enriched with MK-7 (Active Comparator): one study group will receive daily two basic dairy products enriched with MK-7 (50 μg)
  Interventions: Dietary Supplement: basic yogurt enriched with MK-7
- MK-7 containing capsule (Active Comparator): one study group will receive daily a softgel capsule consisting of 50 μg MK-7
  Interventions: Dietary Supplement: MK-7 containing capsule
- nutrient enriched yogurt with MK-7 (Active Comparator): one study group will receive daily two nutrient-enriched dairy products containing extra nutrients and omega-3 FA (fish-oil)
  Interventions: Dietary Supplement: nutrient-enriched yogurt with MK-7

INTERVENTIONS:
Dietary Supplement: MK-7 containing capsule
  Arms: MK-7 containing capsule
Dietary Supplement: basic yogurt enriched with MK-7
  Arms: basic yogurt enriched with MK-7
Dietary Supplement: nutrient-enriched yogurt with MK-7
  Arms: nutrient enriched yogurt with MK-7

SUMMARY:
The objective of this study is to investigate the absorption of menaquinone-7 from a nutrient-enriched dairy product compared to a general dairy product enriched with menaquinone-7 and a menaquinone-7-containing supplement.

DETAILED DESCRIPTION:
In an earlier study, beneficial effects of a nutrient-enriched dairy product on vitamin K-status were observed. The study product contained menaquinone-7 (MK-7) and omega-3 fatty acids for vascular health and extra minerals and antioxidants to support general health. It was the first time that such low dose of MK-7 (50 µg) could significantly improve vascular and general vitamin K-status already after short-term treatment. From the results of this study, it was assumed that the matrix of the dairy product and/or other components in the product, in which the vitamin was offered, contributed to optimal absorption and availability of vitamin K2. In this new study, the uptake and efficacy of MK-7 from the nutrient enriched product is investigated and compared to the uptake and efficacy from a MK-7-containing supplement and a basic dairy product enriched with MK-7.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and postmenopausal women between 45 and 65 years old
* Subjects with body weight and height according to BMI between 20 and 30 kg/m2
* Subjects of Caucasian race
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with hypertension
* Subjects with hypercholesterolemia
* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Subjects with (a history) of diabetes mellitus
* Abuse of drugs and/or alcohol
* Subjects receiving corticosteroid treatment
* Subjects using oral anticoagulants and subjects with clotting disorders
* Subjects using blood pressure-lowering medication
* Subjects using cholesterol-lowering medication
* Subjects using multivitamins or vitamin K supplements
* Subjects consuming high amounts of vitamin K-containing food products
* Subjects with cow's milk allergy and lactose intolerance

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The change in plasma MK-7 concentration after intervention between the three study groups | baseline and 6 weeks

SECONDARY OUTCOMES:
The change in circulating markers of vitamin K-status, undercarboxylated osteocalcin and desphospho-uncarboxylated matrix Gla-protein, after intervention between the three study groups. | baseline and 6 weeks

OTHER OUTCOMES:
The change in circulating vitamin D (25-hydroxy-vitamin D) after intervention between the study groups. | baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK BV Maastricht University
Locations (1):
- VitaK BV / Maastricht University Medical Center, Maastricht, Netherlands